CLINICAL TRIAL: NCT04546009
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of GDC-9545 Combined With Palbociclib Compared With Letrozole Combined With Palbociclib in Patients With Estrogen Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Giredestrant Combined With Palbociclib Compared With Letrozole Combined With Palbociclib in Participants With Estrogen Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer (persevERA Breast Cancer)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO41843; 2020-000119-66 (EudraCT Number); 2023-506911-16-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-08; First posted 2020-09-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Estrogen Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; Letrozole; palbociclib; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Giredestrant + Letrozole-matched Placebo + Palbociclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Letrozole-matched Placebo; Drug: Palbociclib; Drug: LHRH Agonist
- Letrozole + Giredestrant-matched Placebo + Palbociclib (Active Comparator)
  Interventions: Drug: Giredestrant-matched Placebo; Drug: Letrozole; Drug: Palbociclib; Drug: LHRH Agonist

INTERVENTIONS:
Drug: Giredestrant — Giredestrant is taken orally once per day on Days 1-28 of each 28-day treatment cycle.
  Other Names: GDC-9545; RO7197597; RG6171
  Arms: Giredestrant + Letrozole-matched Placebo + Palbociclib
Drug: Giredestrant-matched Placebo — Giredestrant-matched placebo is taken orally once per day on Days 1-28 of each 28-day treatment cycle.
  Arms: Letrozole + Giredestrant-matched Placebo + Palbociclib
Drug: Letrozole — Letrozole 2.5 milligrams (mg) is taken orally once per day on Days 1-28 of each 28-day treatment cycle.
  Arms: Letrozole + Giredestrant-matched Placebo + Palbociclib
Drug: Letrozole-matched Placebo — Letrozole-matched placebo is taken orally once per day on Days 1-28 of each 28-day treatment cycle.
  Arms: Giredestrant + Letrozole-matched Placebo + Palbociclib
Drug: Palbociclib — Palbociclib 125 mg is taken orally once per day on Days 1-21 of each 28-day treatment cycle.
Drug: LHRH Agonist — Only premenopausal/perimenopausal and male participants will receive a luteinizing hormone-releasing hormone (LHRH) agonist on Day 1 of each 28-day treatment cycle. The investigator will determine and supply the appropriate LHRH agonist locally approved for use in breast cancer.

SUMMARY:
This Phase III, randomized, double-blind, placebo-controlled, multicenter study will evaluate the efficacy and safety of giredestrant combined with palbociclib compared with letrozole combined with palbociclib in patients with estrogen receptor (ER)-positive, human epidermal growth factor receptor-2 (HER2)-negative locally advanced (recurrent or progressed) or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* For women who are premenopausal or perimenopausal and for men: treatment with approved LHRH agonist therapy for the duration of study treatment
* Locally advanced (recurrent or progressed) or metastatic adenocarcinoma of the breast, not amenable to treatment with curative intent
* Documented ER-positive tumor and HER2-negative tumor, assessed locally
* Patients who have bilateral breast cancers which are both ER-positive and HER2-negative can be included in the study because the metastases are suitably targeted by the study treatments. If patients have bilateral tumors which are of different biomarker status, then proof of the ER and HER2 status of the metastases is required for study entry
* No history of systemic anti-cancer therapy for locally advanced (recurrent or progressed) or metastatic disease
* Disease recurrence from early-stage breast cancer after standard adjuvant endocrine therapy meeting the protocol-defined criteria of having received at least 24 months of treatment without disease progression during treatment and a disease-free interval since the completion of treatment that was greater than 12 months
* Measurable disease as defined per RECIST v.1.1 or bone only disease which must have at least one predominantly lytic bone lesion confirmed by CT or MRI which can be followed
* Eastern Cooperative Oncology Group Performance Status 0-1
* Adequate organ function

Exclusion Criteria:

* Disease recurrence during or within 12 months of completing prior neoadjuvant or adjuvant treatment with any CDK4/6 inhibitor
* Prior treatment with a selective estrogen receptor degrader (SERD)
* Treatment with any investigational therapy within 28 days prior to study treatment
* Treatment with strong CYP3A inhibitors or inducers within 14 days or 5 drug elimination half-lives (whichever is longer) prior to randomization
* Advanced, symptomatic, visceral spread that is at risk of life-threatening complications in the short term
* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease
* Active cardiac disease or history of cardiac dysfunction, as defined in the protocol
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS), as Determined by the Investigator According to RECIST v1.1 | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 78 months)

SECONDARY OUTCOMES:
Overall Survival | From randomization to death from any cause (up to 78 months)
Objective Response Rate, as Determined by the Investigator According to RECIST v1.1 | From randomization until disease progression or death (up to 78 months)
  The objective response rate is defined as the percentage of participants with a complete response or partial response on two consecutive occasions at least (≥)4 weeks apart.
Duration of Response, as Determined by the Investigator According to RECIST v1.1 | From first occurrence of documented objective response to disease progression or death from any cause, whichever occurs first (up to 78 months)
Clinical Benefit Rate, as Determined by the Investigator According to RECIST v1.1 | From randomization until disease progression or death (up to 78 months)
  The clinical benefit rate is defined as the percentage of participants with stable disease for ≥24 weeks or a complete response or partial response.
Time to Confirmed Deterioration in Pain Level, Defined as the Time to First Documented ≥2-Point Increase from Baseline in the 'Worst Pain' Item from the Brief Pain Inventory-Short Form (BPI-SF) Questionnaire | From Baseline until treatment discontinuation (up to 78 months)
Time to Confirmed Deterioration in Pain Presence and Interference, Defined as the Time to First Documented ≥10-Point Increase from Baseline in the EORTC QLQ-C30 Linearly Transformed Pain Scale Score | From Baseline until treatment discontinuation (up to 78 months)
  EORTC QLQ-C30 = European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire
Time to Confirmed Deterioration in Physical Functioning, Defined as the Time to First Documented ≥10-Point Decrease from Baseline in the EORTC QLQ-C30 Linearly Transformed Physical Functioning Scale Score | From Baseline until treatment discontinuation (up to 78 months)
Time to Confirmed Deterioration in Role Functioning, Defined as the Time to First Documented ≥10-Point Decrease from Baseline in the EORTC QLQ-C30 Linearly Transformed Role Functioning Scale Score | From Baseline until treatment discontinuation (up to 78 months)
Time to Confirmed Deterioration in Global Health Status and Quality of Life (GHS/QoL), Defined as the Time to First Documented ≥10-Point Decrease from Baseline in the EORTC QLQ-C30 Linearly Transformed GHS/QoL Scale Score | From Baseline until treatment discontinuation (up to 78 months)
Number of Participants with Adverse Events, Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v5.0) | From treatment initiation until 30 days after the final dose of study treatment (up to 78 months)
Number of Participants with Vital Sign Abnormalities Over the Course of the Study | Baseline, Days 1 and 15 of Cycles 1 and 2, and Day 1 of each cycle thereafter until treatment discontinuation (1 cycle is 28 days)
  Vital signs include respiratory rate, pulse rate, and systolic and diastolic blood pressure while the participant is in a seated position, and temperature.
Plasma Concentration of Giredestrant at Specified Timepoints | Days 1 and 15 of Cycle 1; Day 1 of Cycles 2, 4, 8, and 16 (1 cycle is 28 days)
Plasma Concentration of Palbociclib at Specified Timepoints | Days 1 and 15 of Cycle 1 (1 cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (255):
- United States (37):
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Kaiser Permanente - San Leandro Medical Center, San Leandro, California
  - Stanford Univ Medical Center, Stanford, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Florida Cancer Specialists - Fort Myers (Broadway), Fort Myers, Florida
  - Memorial Regional Cancer Ctr, Hollywood, Florida
  - University of Miami, Miami, Florida
  - SCRI Florida Cancer Specialists North, St. Petersburg, Florida
  - SCRI Florida Cancer Specialists PAN, Tallahassee, Florida
  - Kaiser Permanente - Moanalua Medical Center, Honolulu, Hawaii
  - Mercy Medical Center, Baltimore, Maryland
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - HCA Midwest Division, Kansas City, Missouri
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Astera Cancer Care East Brunswick, East Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center at Bergen, Montvale, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - MSKCC @ Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Providence Portland Medical Ctr, Portland, Oregon
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - DFW, Dallas, Texas
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (7):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital de Onc Angel Roffo, Buenos Aires
  - Organización medica de Investi, Cap Fed
  - Hospital Britanico, Ciudad Autonoma Bs As
  - Hospital Provincial del Centenario, Rosario
  - Instituto de Oncología de Rosario, Rosario
  - CEMER Centro Medico de Enfermedades Respiratorias, Vicente López
- Australia (6):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fiona Stanley Hospital - Medical Oncology, Murdoch, Western Australia
- Austria (3):
  - Uniklinikum Salzburg, LKH, Salzburg
  - A.Ö. LHK, Steyr
  - Medizinische Universität Wien, Vienna
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - Jessa Zkh (Campus Virga Jesse), Hasselt
- Brazil (8):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
  - Beneficencia Portuguesa de Sao Paulo, São Paulo, São Paulo
- Canada (11):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - BC Cancer ? Surrey, Surrey, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health System Brampton Civic Hospital, Brampton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Universite de Montreal - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l?Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- China (17):
  - Anyang Tumor Hosptial, Anyang
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Cancer Hospital, Beijing
  - the First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Fujian Medical University Union Hospital, Fujian
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Shengjing Hospital of China Medical University, Shenyang
  - Liaoning cancer Hospital & Institute, Shenyang
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
- Denmark (3):
  - Herlev Hospital, Herlev
  - Sjællands Universitetshospital, Næstved, Næstved
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
- France (9):
  - ICO Paul Papin, Angers
  - Centre Hospitalier de La Cote Basque, Bayonne
  - Chd de Vendee, La Roche-sur-Yon
  - Institut régional du Cancer Montpellier, Montpellier
  - Chu La Miletrie, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - ICL, Saint-Priest-en-Jarez
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (19):
  - Ambulantes Tumorzentrum Spandau, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg GmbH, Georgsmarienhütte
  - Dres.Andreas Ammon und Dirk Meyer, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Facharztzentrum Eppendorf, Studien GbR, Hamburg
  - Medizinische Hochschule Zentrum Frauenheilkunde Abt.Gynäkologische Onkologie, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Praxis Köppler, Heymann, Weide, Thomalla, Koblenz
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - St. Elisabeth-Krankenhaus, Senologie/Brustzentrum, Leipzig
  - Universitätsklinikum Mannheim, Mannheim
  - Klinik & Poliklinik für Frauenheilkunde und Geburtshilfe, Campus Innenstadt, München
  - MVZ für Hämatologie und Onkologie Ravensburg GmBH, Ravensburg
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH, Trier
  - Dres. Helmut Forstbauer, Carsten Ziske und Kollegen, Troisdorf
  - Universitätsklinik Tübingen, Tübingen
- Greece (4):
  - Anticancer Hospital Ag Savas, Athens
  - Anticancer Hospital Ag. Savas, Athens
  - Euromedical General Clinic of Thessaloniki, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (2):
  - Honvédelmi Minisztérium Állami Egészségügyi Központ;Onkológiai Osztály, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
- Israel (3):
  - Davidof Center - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Ctr, Tel Aviv
- Italy (11):
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - IRCCS Istituto Regina Elena (IFO), Rome, Lazio
  - Az. Osp. Spedali Civili, Brescia, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Asst Di Monza, Monza, Lombardy
  - Humanitas Centro Catanese Di Oncologia, Misterbianco (CT), Sicily
  - Fondazione del Piemonte per l?Oncologia (IRCCS), Candiolo, Trentino-Alto Adige
  - Ospedale Civile - Livorno, Livorno, Tuscany
  - Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
  - Azienda ULSS 8 Berica, Vicenza, Veneto
- Japan (22):
  - Nagoya University Hospital, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Hyogo Cancer Center, Hyōgo
  - University of Tsukuba Hospital, Ibaraki
  - Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Fukushima Medical University Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Naha-nishi Clinic, Okinawa
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Showa Medical University Hospital, Tokyo
- Mexico (7):
  - Health Pharma Professional Research, CD Mexico, Mexico CITY (federal District)
  - Centro de Atencion Oncologica Viva S de RL de CV, Mexico City, Mexico CITY (federal District)
  - Filios Alta Medicina, Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Morelia
  - Sociedad de Metabolismo y Corazón (SOMECO), Veracruz
- Auckland City Hospital, Auckland, New Zealand
- Peru (4):
  - Oncosalud Sac, Lima
  - Instituto Peruano de Oncología y Radioterapia, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Instituto Regional de Enfermedades Neoplasicas - IREN Norte, Trujillo
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Szpital Morski im. PCK, Gdynia
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad, Warsaw
- Portugal (4):
  - IPO de Coimbra, Coimbra
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
  - IPO do Porto, Porto
- Russia (7):
  - SBIH "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of DHM", Moskva, Moscow Oblast
  - Podolsk City Clinical Hospital, Podolsk, Moscow Oblast
  - Respublikanskiy Onkologicheskiy Dispanser, Saransk, Respublika Mordoviya
  - Ryazan Regional clinical oncology dispensary, Ryazan, Ryazan Oblast
  - GBUZ Saint Petersburg Clinical Research Center of Specialized Types of Care (Oncology), Saint Petersburg, Sankt-Peterburg
  - Chelyabinsk region oncology dispensary, Chelyabinsk
  - Multidisciplinary clinic Reaviz, Samara
- South Korea (13):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (15):
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Centro Oncologico MD Anderson Internacional, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - HM Sanchinarro ? CIOCC, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (6):
  - China Medical University Hospital, Taichung
  - National Cheng Kung Uni Hospital, Tainan
  - Veterans General Hospital, Taipei
  - National Taiwan Uni Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hosipital at Linkou, Taoyuan Hsien
- Thailand (5):
  - Chulalongkorn Hospital, Faculty of Medicine, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hosp, Chang Mai
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (8):
  - Hacettepe Uni Medical Faculty Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Medipol University Medical Faculty, Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Kocaeli University Faculty of Medicine, İzmit
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
  - 19 Mayis University Medical Faculty, Samsun
- Ukraine (5):
  - Municipal Institution City Clinical Hospital #4 of Dnipro City Council, Dnipropetrovsk, Katerynoslav Governorate
  - SI Institute of general&urgent surgery n/a Zaytseva V.T NAMSU, Kharkiv, Kharkiv Governorate
  - Ivano-Frankivsk Regional Oncology Center, Ivano-Frankivsk
  - ME Kryviy Rih Oncology Dispensary of Dnipropetrovs?k Regional Council, Kryvyi Rih
  - Sumy Regional Clinical Onc Ctr, Sumy
- United Kingdom (10):
  - Royal Sussex County Hospital, Brighton
  - Leicester Royal Infirmary, Leicester
  - University College London Hospital, London
  - Royal Free Hospital, London
  - Guys & St Thomas Hospital, London
  - Maidstone Hospital, Maidstone
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital, Plymouth
  - Royal Marsden Hosp NHS Fnd, Sutton
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing